CLINICAL TRIAL: NCT07005193
Title: Effects of Liquefied Petroleum Gas and Ventilation Interventions on Reducing Household Air Pollution From Solid Fuel Use and Improving Cardiopulmonary Health: A Multi-center, 2×2 Factorial Randomized Controlled Trial
Brief Title: Effects of LPG and Ventilation Interventions on Reducing HAP and Improving Cardiopulmonary Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Kuai Yu, Associate Research Fellow, Principal Investigator, Huazhong University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2023ZD0509900
Record Dates: First submitted 2025-05-08; First posted 2025-06-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiopulmonary Function; Environmental Exposures
MeSH Terms: interventions — Cooking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Solid fuel + no ventilation (control). (No Intervention): Solid fuel + no ventilation facilities group: Continued use of solid fuels without ventilation facilities, with a one-time financial compensation provided post-intervention.
- B: LPG + no ventilation. (Experimental): Liquefied petroleum gas (LPG) + no ventilation facilities group: Provided with LPG stoves and instructed to use them for cooking, with regular LPG supply during the intervention period.
  Interventions: Behavioral: Using liquefied gas for cooking
- C: Solid fuel + ventilation. (Experimental): Solid fuel + ventilation facilities group: Maintained solid fuel usage habits while provided with ventilation facilities and instructed to use them during cooking, with electricity costs compensated during the intervention.
  Interventions: Device: Using rang hood during cooking
- D: LPG + ventilation. (Experimental): LPG + ventilation facilities group: Provided with both LPG stoves and ventilation facilities, instructed to use both during cooking, with regular LPG supply and electricity cost compensation throughout the intervention period.
  Interventions: Device: Using rang hood during cooking; Behavioral: Using liquefied gas for cooking

INTERVENTIONS:
Device: Using rang hood during cooking — Cooking ventilation facilities
  Arms: C: Solid fuel + ventilation.; D: LPG + ventilation.
Behavioral: Using liquefied gas for cooking — Using liquefied gas instead of solid fuels for cooking
  Arms: B: LPG + no ventilation.; D: LPG + ventilation.

SUMMARY:
The goal of this clinical trial is to evaluate the independent and synergistic effects of liquefied petroleum gas (LPG) substitution and improved ventilation on household air pollution (HAP) reduction and cardiopulmonary health. The main questions it aims to answer are:

1. Does LPG substitution or improved ventilation reduce HAP and improve cardiopulmonary health?
2. Would the combined intervention of LPG substitution and improved ventilation outperform single interventions?
3. What is the cost-effectiveness of such interventions, and are they sustainable?

Participants will be randomized in 4 groups:

A: Solid fuel + no ventilation facilities group (195 households): Continued use of solid fuels without ventilation facilities, with a one-time financial compensation provided post-intervention; B: Liquefied petroleum gas (LPG) + no ventilation facilities group (195 households): Provided with LPG stoves and instructed to use them for cooking, with regular LPG supply during the intervention period; C: Solid fuel + ventilation facilities group (195 households): Maintained solid fuel usage habits while provided with ventilation facilities and instructed to use them during cooking, with electricity costs compensated during the intervention; D: LPG + ventilation facilities group (195 households): Provided with both LPG stoves and ventilation facilities, instructed to use both during cooking, with regular LPG supply and electricity cost compensation throughout the intervention period.

ELIGIBILITY:
1. Inclusion Criteria Primary Participants：

   * Primary use of solid fuels (coal, wood, charcoal, or crop residues) for cooking;
   * Kitchen is suitable for installing ventilation facilities;
   * The main cook in the household (cooking frequency ≥5 times/week);
   * Aged between 18 and 74 years;
   * Local permanent residents with no plans for long-term travel or relocation within one year.

   Secondary Participants

   ● Elderly individuals aged 65-74 who lived with the included primary participants.
2. Exclusion Criteria:

   * Clinical diagnosis of major chronic diseases such as severe respiratory diseases, cardiovascular diseases, malignant tumors, or end-stage renal disease;
   * Pregnant or breastfeeding women;
   * Current smokers or individuals with self-reported exposure to productive dust or other occupational hazards;
   * Individuals who are unable to fully understand the study process or clearly express their own complaints, such as those with psychiatric disorders or severe neuroses, or who cannot cooperate with the study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Number of Ultrafine particles (UFP) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: particles/cm³, Measuring instrument: TSI NanoScan (TSI, USA), MicroPEM (PennEngineering, USA), Gillian5000 (Sensidyne, USA), Measurement method: Monitoring device sensors.
Change in the Concentrations of PM2.5 | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: TSI NanoScan (TSI, USA), MicroPEM (PennEngineering, USA), Gillian5000 (Sensidyne, USA), Bbair (Yuanrui Environmental Protection Technology Co., Ltd, China) , Measurement method: Monitoring device sensors.
Change in the Heart Rate Variability (HRV) Measured by 12-lead ECG | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Heart rate variability measured using standard 12-lead electrocardiogram (ECG). Measuring instrument: HeaLink heart rate sensor (Henan Link Medical Technology Co., Ltd., China), The time-domain indicators include:SDNN: Standard deviation of all normal-to-normal (NN) intervals over 24 hours / SDANN: Standard deviation of the average NN intervals calculated over 5-minute segments throughout 24 hours / RMSSD: Root mean square of successive differences between adjacent NN intervals over 24 hours.
  The frequency-domain indicators include: TP: Total power / LF: Low-frequency power / HF: High-frequency power / LF/HF: Ratio of low-frequency to high-frequency power.
Change in the Forced Vital Capacity (FVC) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Forced Vital Capacity measured using spirometer (HI105; Chestgraph, Japan). Units of Measure: Liters. Method of Measurement: Standardized spirometric testing protocol.
Change in the Forced Expiratory Volume in 1 Second (FEV1) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Forced Expiratory Volume in 1 Second measured using spirometer (HI105; Chestgraph, Japan). Units of Measure: Liters. Method of Measurement: Standardized spirometric testing protocol.

SECONDARY OUTCOMES:
Change in the Concentrations of Specific Chemical Components in Particulate Matter | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: Gilian (Sensidyne, USA), PEM-2-2.5 (MSP,USA), Measurement method: ICP-MS (Inductively Coupled Plasma Mass Spectrometry) and GC-MS/MS (Gas Chromatography-Tandem Mass Spectrometry).
Change in the Concentrations of Ozone (O₃) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: AEROQUAL Series 500 (Aeroqual, New Zealand), Measurement method: Monitoring device sensors.
Change in the Concentrations of Black Carbon (BC) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: Model AE51 (AethLabs, USA), Measurement method: Monitoring device sensors.
Change in the Systolic and Diastolic Blood Pressure | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: mmHg, Instrument: Omron (Japan);
Change in the Fractional Exhaled Nitric Oxide (FeNO) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ppb , Instrument: NIOX VERO (Aerocrine AB; Solna, Sweden);
Change in the Pulse Wave Velocity (PWV) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Assessed using an arterial stiffness analyzer (Itamar Medical, Israel) to measure arterial stiffness in meters per second (m/s).
Change in the Forced Expiratory Flow at 75% of FVC (FEF75) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Forced Expiratory Flow at 75% of Forced Vital Capacity measured in Liters/Second. Units of Measure: Liters/Second. Method of Measurement: Standardized spirometric testing protocol.
Change in the Forced Expiratory Flow at 50% of FVC (FEF50) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Forced Expiratory Flow at 50% of Forced Vital Capacity measured in Liters/Second. Units of Measure: Liters/Second. Method of Measurement: Standardized spirometric testing protocol.
Change in the Forced Expiratory Flow at 25% of FVC (FEF25) | 1 year, with follow-ups at 6, 1 protocol.2, 24, and 36 months
  Forced Expiratory Flow at 25% of Forced Vital Capacity measured in Liters/Second. Method of Measurement: Standardized spirometric testing
Change in the Peak Expiratory Flow (PEF) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Peak Expiratory Flow measured using spirometer (HI105; Chestgraph, Japan).Units of Measure: Liters/Second. Method of Measurement: Standardized spirometric testing protocol.
Change in the Cardio-Ankle Vascular Index (CAVI) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Measured using arterial stiffness analyzer (Itamar Medical, Israel) to assess arterial stiffness.
Change in the Peripheral Arterial Tone (PAT) Index | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Assessed using the EndoPAT noninvasive endothelial function detection system (Itamar Medical, Israel).
Change in the Environmental Noise Level | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: dB, Measuring instrument: Model ASV5910+ (Aihua Instruments Co., Ltd, China) , Measurement method: Monitoring device sensors.
Change in the Concentrations of Internal Exposure to PAHs and VOCs | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ng/mL, Measuring samples: Urine samples, Measurement method: GC-MS/MS.
Change in the Concentrations of Internal Exposure to Metal Elements | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ng/mL, Measuring samples: Blood and urine samples, Measurement method: ICP-MS.
Change in the Concentrations of Total Volatile Organic Compounds (TVOCs) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: Model TG-503 (GrayWolf, USA), Measurement method: Monitoring device sensors
Change in the Concentrations of Nitrogen Dioxide (NO₂) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: AEROQUAL Series 500 (Aeroqual, New Zealand) , Measurement method: Monitoring device sensors.
Change in the Concentrations of PM1 / PM10 | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Unit: ug/m3, Measuring instrument: TSI NanoScan (TSI, USA), MicroPEM (PennEngineering, USA), Gillian5000 (Sensidyne, USA), Bbair (Yuanrui Environmental Protection Technology Co., Ltd, China) , Measurement method: Monitoring device sensors.

OTHER OUTCOMES:
Change in the Serum Levels of Myocardial Function Biomarkers (BNP, NT-proBNP, Follistatin, Myoglobin, CK-MB, Troponin I, Troponin T) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Units (e.g., pg/mL or ng/mL) depend on the specific analyte and assay standard. Serum concentrations of the following myocardial function biomarkers will be measured: B-type Natriuretic Peptide (BNP), N-terminal prohormone BNP (NT-proBNP) , Follistatin, Myoglobin, Creatine Kinase-MB (CK-MB), Troponin I, Troponin T, Method: MILLIPLEX: serum;
Change in the Serum Levels of Club Cell Protein 16 (CC16) and Surfactant Protein D (SP-D) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Lung epithelial injury will be assessed by measuring serum levels of:Club Cell Protein 16 (CC16), Surfactant Protein D (SP-D). Method: enzyme-linked immunosorbent assay (ELISA) in serum samples. Units are typically pg/mL or ng/mL, depending on assay specifications.
Change in the Serum Levels of Blood Glucose, Insulin, and C-Peptide | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Method: glucose oxidase method: serum. Units (e.g., mmol/L for glucose, μIU/mL or pmol/L for insulin and C-peptide) depend on assay specifications
Change in the Genome-wide DNA Methylation Levels in Blood Samples | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Epigenetic alterations will be assessed by measuring genome-wide DNA methylation levels using peripheral blood-derived DNA.
Change in the Serum Levels of Oxidative Stress Biomarkers | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Oxidative stress status will be assessed by measuring serum concentrations of the following biomarkers using ELISA assays: Angiotensin II (Ang-II) / NADPH oxidase (NOX) / Superoxide dismutase (SOD) / Glutathione (GSH) / Malondialdehyde (MDA) / Oxidized low-density lipoprotein (ox-LDL).
Change in the Serum Levels of HPA Axis Stress Hormones (Cortisol, ACTH, CRH) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  The hypothalamic-pituitary-adrenal (HPA) axis function will be evaluated by measuring serum concentrations of: Cortisol / Adrenocorticotropic hormone (ACTH) / Corticotropin-releasing hormone (CRH). Measurements will be performed using enzyme-linked immunosorbent assay (ELISA).
Change in the Concentrations of Plasma Triacylglycerols (TAG) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 40 triacylglycerols in plasma assessed using LC-MS.Units of Measure: ng/mL
Change in the Concentrations of Plasma Diglycerides (DAG) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 4 diglycerides in plasma measured using LC-MS-based metabolomics. Units of Measure: ng/mL
Change in the Concentrations of Plasma Cholesteryl Esters (CE) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 14 cholesteryl esters in plasma determined using targeted LC-MS. Units of Measure: ng/mL
Change in the Concentrations of Plasma Phosphatidylethanolamines (PE) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 11 PE species in plasma determined using LC-MS-based metabolomics. Units of Measure: ng/mL
Change in the Concentrations of Plasma Lysophosphatidylethanolamines (LPE) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 4 LPE species in plasma assessed using LC-MS. Units of Measure: ng/mL
Change in the Concentrations of Plasma Sphingomyelins (SM) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 20 sphingomyelins in plasma measured using LC-MS-based metabolomics. Units of Measure: ng/mL
Change in the Concentrations of Plasma Phosphatidylcholines (PC) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 50 phosphatidylcholines in plasma measured using LC-MS-based targeted metabolomics. Units of Measure: ng/mL
Change in the Concentrations of Plasma Lysophosphatidylcholines (LPC) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 18 lysophosphatidylcholines in plasma determined using LC-MS metabolomic analysis. Units of Measure: ng/mL
Change in the Concentrations of Plasma Ceramides | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 5 ceramides (Cer) in plasma measured by targeted LC-MS metabolomics. Units of Measure: ng/mL
Change in the Concentrations of Other Polar Small Molecule Metabolites in Plasma | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 14 other polar metabolites measured in plasma using LC-MS-based targeted metabolomics. Units of Measure: μmol/L
Change in the Concentrations of Plasma Carnitines and Acylcarnitines | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 12 carnitines and acylcarnitines measured in plasma using LC-MS. Units of Measure: μmol/L
Change in the Concentrations of Plasma Amino Acids | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentrations of 26 amino acids measured in plasma using targeted LC-MS metabolomics. Units of Measure: μmol/L
Change in the Concentrations of Tissue Plasminogen Activator (t-PA) in Serum | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentration of t-PA in serum measured using ELISA assay. Units of Measure: ng/mL
Change in the Concentrations of Plasminogen Activator Inhibitor-1 (PAI-1) in Serum | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentration of PAI-1 in serum measured using ELISA assay. Units of Measure: ng/mL
Change in the Concentrations of D-dimer in Serum | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentration of D-dimer in serum measured using ELISA assay. Units of Measure: ng/mL
Change in the Concentrations of Fibrinogen in Serum | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentration of fibrinogen in serum measured using ELISA assay. Units of Measure: mg/dL
Change in the Concentrations of Von Willebrand Factor (vWF) in Serum | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentration of Von Willebrand factor (vWF) measured in serum using ELISA assay. Units of Measure: μg/mL
Change in the Concentrations of Soluble CD40 Ligand (sCD40L) in Serum | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Concentration of soluble CD40 ligand (sCD40L) measured in serum using ELISA assay. Units of Measure: ng/mL
Change in the Mean Platelet Volume (MPV) (fL) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Average size of platelets measured in the blood. Units of Measure: fL. Method of Measurement: Clinical laboratory testing.
Change in the Platelet Distribution Width (PDW) (%) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Measurement of variability in platelet size. Units of Measure: fL. Method of Measurement: Clinical laboratory testing
Change in the Red Cell Distribution Width - Coefficient of Variation (RDW-CV) (%) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  RDW-CV reflects relative size variability among red blood cells. Units of Measure: %. Method of Measurement: Clinical laboratory testing
Change in the Red Cell Distribution Width - Standard Deviation (RDW-SD) (fL) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  RDW-SD reflects variation in red cell size. Units of Measure: fL. Method of Measurement: Clinical laboratory testing.
Change in the Platelet Count (PLT) (10⁹/L) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Platelet count measured from plasma samples. Units of Measure: 10⁹/L. Method of Measurement: Clinical laboratory testing.
Change in the Mean Corpuscular Hemoglobin Concentration (MCHC) (g/dL) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Mean concentration of hemoglobin in red blood cells. Units of Measure: g/dL. Method of Measurement: Clinical laboratory testing
Change in the Mean Corpuscular Hemoglobin (MCH) (pg/cell) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Mean corpuscular hemoglobin value measured in plasma. Units of Measure: pg (picograms). Method of Measurement: Clinical laboratory testing
Change in the Mean Corpuscular Volume (MCV) (fL) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Mean corpuscular volume assessed from plasma samples. Units of Measure: fL (femtoliters). Method of Measurement: Clinical laboratory testing
Change in the Hematocrit (HCT) Level (%) | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Hematocrit percentage measured from plasma samples.Units of Measure: %. Method of Measurement: Clinical laboratory testing
Change in the Concentration of Hemoglobin Concentration (HGB) in Plasma | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Hemoglobin concentration in plasma measured in clinical laboratory. Units of Measure: g/dL. Method of Measurement: Clinical laboratory testing.
Change in the Concentration of Red Blood Cells (RBC) in Plasma | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Red blood cell count measured from plasma samples using automated hematology analyzer.Units of Measure: 10¹²/L. Method of Measurement: Clinical laboratory testing.
Change in the Concentration of White Blood Cells (WBC) in Plasma | 1 year, with follow-ups at 6, 12, 24, and 36 months
  White blood cell count measured from plasma samples using automated hematology analyzer. Units of Measure: 10⁹/L. Method of Measurement: Clinical laboratory testing.
Change in the Sleep Parameters Measured by ActiGraph GT3X-BT | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Objective sleep characteristics-including total sleep time, sleep efficiency, sleep latency, and wake after sleep onset-will be measured using the ActiGraph GT3X-BT wearable device. Units of Measure: Minutes for time-based parameters; percent for sleep efficiency.
Change in the Pittsburgh Sleep Quality Index (PSQI) Score | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-reported questionnaire. Units of Measure: Points on a scale.
Change in the Serum Levels of Systemic Inflammatory Cytokines and Biomarkers | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Systemic inflammation will be assessed by measuring serum concentrations of multiple cytokines and biomarkers using the MILLIPLEX multiplex assay platform. Included analytes are: C-reactive protein (CRP) / Interleukins: IL-1β, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-17A / Macrophage-Derived Chemokine (MDC) / Tumor Necrosis Factor-alpha (TNF-α) / Interferon-gamma (IFN-γ) / Monocyte Chemoattractant Protein-1 (MCP-1). Units are typically pg/mL.
Change in the Expression Levels of mRNAs and miRNAs in Blood and Plasma | 1 year, with follow-ups at 6, 12, 24, and 36 months
  Transcriptomic profiling will be performed to measure the expression levels of mRNAs and microRNAs (miRNAs) in blood and plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kuai Yu, Principal Investigator — Huazhong University of Science and Technology
Locations (3):
- China (3):
  - Suiping County Health Center, Zhumadian, Henan
  - Hong'an County Health Center, Huanggang, Hubei
  - Longhui County Health Center, Shaoyang, Hunan